CLINICAL TRIAL: NCT04883372
Title: Assessment of the Impact of Telemedicine in Insulin-dependent Diabetic Patients Through the ETAPES Program.
Brief Title: Study of the Effect of Telemedicine on Glycemic Control for Patients With Diabetes and Treated With Insulin
Acronym: TLS-DIAB
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/0013
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Diabetes
Keywords: Telemedicine; telemonitoring; diabetes; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: continuous glucose monitoring — a continuous glucose monitoring CGM system through the ETAPES telemedicine program

SUMMARY:
The purpose of this study is to assess glycemic control changes in insulin-treated patients with diabetes using a continuous glucose monitoring CGM system through the ETAPES telemedicine program.

DETAILED DESCRIPTION:
Diabetes is currently one of the major health challenges. According to the International Diabetes Federation (IDF), the number of people with diabetes has tripled in the last 20 years and will reach 463 million cases in 2020. This chronic disease causes degenerative complications that affect the quality of life of patients and increase the morbidity and mortality rate. This is due to limited access to health professionals, inadequate patient education and especially poor self-management of their disease which hinders adequate glycemic control of diabetes. The daily routine of a type 1 diabetic patient includes self-monitoring of blood glucose levels as well as several insulin injections per day or the use of an insulin pump. However, this treatment does not prevent the occurrence of micro and/or macroangiopathic complications, especially when the diabetes is poorly controlled. Therefore, optimal and large-scale glycemic control can have a significant clinical, social and economic impact. The Diabetes Control and Complications Trial (DCCT) has shown that intensive glycemic control delays or prevents the occurrence of microvascular and macrovascular complications. Intensive treatment, education and support for diabetes self-management improves glycated hemoglobin levels, reducing the risk of developing degenerative complications. This is accompanied by a positive psychosocial and behavioral effect. It is in this context that telemedicine, via remote monitoring, can improve glycemic control. Diabetes remains one of the most suitable specialties for telemedicine, especially with the advent of continuous glucose measurements reimbursed by health insurance since 2017.

Since the 1990s, several telemonitoring projects have demonstrated the value of constant support for diabetic patients, resulting in a significant improvement in HbA1c; the patient becomes an actor in his or her management, with better appropriation of the disease and better compliance. Remote monitoring is one of the 5 telemedicine procedures defined in France. It allows a medical professional to remotely interpret the data necessary for a patient's medical follow-up and to make decisions regarding the patient's care.

The French health authorities have set up national experiments on remote monitoring of diabetes under real conditions, such as the ETAPES program, whose objective is to evaluate the clinical, medico-economic and quality of life benefits of patients who benefit from remote monitoring. This program has 3 components: remote medical monitoring of patients including remote interpretation of patient results and adaptation of treatment, therapeutic support through face-to-face or remote sessions and the use of a remote monitoring platform that provides the link between the patient and the medical team.

In December 2019, the endocrinology department of the CHSF decided to implement the ETAPES program via the LIBREVIEW technical solution in order to better support unbalanced insulin-treated diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

For people with T1D, inclusion criteria in the ETAPES program were:

* new onset diabetes (< 6 months) or diabetes duration > 6 months with HbA1C ≥ 8% twice over the last 6 months in people aged over 18 years
* new onset diabetes (< 6 months) or diabetes duration > 6 months with HbA1C ≥ 8.5% twice over the last 6 months in people aged between 12 and 17 years.

For people with T2D, inclusion criteria were diabetes duration > 12 months with HbA1C ≥ 9% twice over the last 6 months in people aged over 18 years.

Exclusion Criteria:

* patients objecting to research

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: insulin-treated diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
glycated hemoglobin | at 3 months
  glycated hemoglobin
glycated hemoglobin | at 6 months
  glycated hemoglobin

SECONDARY OUTCOMES:
glycated hemoglobin | at 3 months
  time spent in the target
glycated hemoglobin | at 6 months
  time spent in the target
Time above target (TAR) | at 3 months
  Change in time above target (TAR) of hyperglycemia, > 250 mg/dL, from 181 to 250 mg/dL
Time above target (TAR) | at 6 months
  Change in time above target (TAR) of hyperglycemia, > 250 mg/dL, from 181 to 250 mg/dL
Time spent below target (TBR) | at 3 months
  Change in time spent below target (TBR) of hypoglycemia from 54 to 69 mg/dL and < 54 mg/dL
Time spent below target (TBR) | at 6 months
  Change in time spent below target (TBR) of hypoglycemia from 54 to 69 mg/dL and < 54 mg/dL

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No